CLINICAL TRIAL: NCT05738655
Title: Effectiveness of Pumpkin Seed Extract on Improving Blood Sugar Level in Subhealth Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Greenyn Biotechnology Co., Ltd. (Industry)
Collaborators: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A-111-110
Record Dates: First submitted 2023-02-01; First posted 2023-02-22 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Diabetes; Metabolic Disease
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Placebo capsule, one capsule/day (300 mg/day) for 3 months
  Interventions: Dietary Supplement: Placebo
- Low dose (Experimental): Pumpkin seed extract capsule, one capsule/day (300 mg/day) for 3 months
  Interventions: Dietary Supplement: Pumpkin seed extract (Low dose)
- High dose (Experimental): Pumpkin seed extract capsule, two capsules/day (600 mg/day) for 3 months
  Interventions: Dietary Supplement: Pumpkin seed extract (High dose)

INTERVENTIONS:
Dietary Supplement: Pumpkin seed extract (Low dose) — Pumpkin seed extract standardized with specific peptides (300 mg/day)
  Arms: Low dose
Dietary Supplement: Pumpkin seed extract (High dose) — Pumpkin seed extract standardized with specific peptides (600 mg/day)
  Arms: High dose
Dietary Supplement: Placebo — Placeo (300 mg/day)
  Arms: Placebo group

SUMMARY:
This randomized, double-blind, placebo-controlled, and parallel clinical study aims to investigate the effectivness of a pumpkin seed extract on blood sugar management in subhealth people.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood sugar levels from 100 to 125 mg/dL
* Glycated hemoglobin levels from 5.7 to 6.4%
* 2-hour OGTT levels from 140 to 199 mg/dL

Exclusion Criteria:

* Pregnant women or preparing for pregnancy.
* Lactating women.
* Women gave birth 6 months before the study.
* Poor kindy funciton
* Severe cardiovascular or other chronic diseases
* Patients with type I or II diabetes
* Poor compliance
* Alcohol abuser
* Using anti-diabetic or weight managent supplements
* Blood transfusion three months before the study
* Pumpkin seed allergy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical analysis | Baseline up to 12 weeks
  Changes in fasting blodd sugar levels of 60 pariticpants will be analyzed between baseline and week 12.
Biochemical analysis | Baseline up to 12 weeks
  Changes in glycosylated hemoglobin levels of 60 pariticpants will be analyzed between baseline and week 12.
Biochemical analysis | Baseline up to 12 weeks
  Changes in insulin levels of 60 pariticpants will be analyzed between baseline and week 12.
Biochemical analysis | Baseline up to 12 weeks
  Changes in incremental area under the curve for glucose for 60 pariticpants will be analyzed between baseline and week 12.
Hormone analysis | Baseline up to 12 weeks
  Changes in GLP-1 levels of 60 pariticpants will be analyzed between baseline and week 12.
Hormone analysis | Baseline up to 12 weeks
  Changes in DPP4 levels of 60 pariticpants will be analyzed between baseline and week 12.
Hormone analysis | Baseline up to 12 weeks
  Changes in adiponectin levels of 60 pariticpants will be analyzed between baseline and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shun Wu, MD, Principal Investigator — WanFang Hospital
Locations (1):
- WanFang Hospital, Taipei, Taiwan